CLINICAL TRIAL: NCT04106817
Title: A Phase I, Open-label, Ascending Dose Study to Determine the Safety and Reactogenicity of a Wild Type Seasonal A/California/ H1N1 2009 Influenza Challenge Virus in Healthy Volunteers, Following a Single Intranasal Administration
Brief Title: Single Ascending Dose Challenge Study to Determine Safety and Reactogenicity of an Influenza Challenge Virus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: WCCT Global (Industry)
Collaborators: Stanford University (Other); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: WCCTG 14-01
Record Dates: First submitted 2019-09-24; First posted 2019-09-27 (Actual); Results first posted 2019-11-19 (Actual); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Experimental): 1:10 dilution of neat virus (0.25mL of 1:10 dilution per nostril of neat virus; approximate quantity 3.5 x 10^6TCID50/dose)
  Interventions: Biological: Live, wild-type A/California/H1N1 2009 influenza virus
- Cohort 2 (Experimental): 1:5 dilution of neat virus (0.25mL of 1:5 dilution per nostril of neat virus; approximate quantity 7 x 10^6TCID50/dose)
  Interventions: Biological: Live, wild-type A/California/H1N1 2009 influenza virus
- Cohort 3 (Experimental): 1:10 dilution of neat virus (0.5mL of 1:10 dilution per nostril of neat virus; approximate quantity 7 x 10^6TCID50/dose)
  Interventions: Biological: Live, wild-type A/California/H1N1 2009 influenza virus

INTERVENTIONS:
Biological: Live, wild-type A/California/H1N1 2009 influenza virus — Live, wild type influenza A virus that was inoculated and manufactured in allantoic fluid of SPF embryonated hen eggs

SUMMARY:
This is a non-controlled, open-label, single-center, dose-escalation study to determine the safety, infectivity, and immune responses elicited from of the potential influenza virus challenge strain. The study objective is to determine the dose with the optimal safety profile and infectivity rate of the viral challenge strain in healthy volunteers for use in subsequent challenge intervention studies to test potential influenza vaccines and/or therapeutics.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, as determined by medical history, physical examination, vital signs, echocardiogram, 12-lead ECG, and clinical safety laboratory examinations at baseline, as determined by the Investigator.
* Absent or low levels of detectable pre-existing antibodies to influenza virus subtypes, including as a minimum the challenge strain, as determined by an HAI titer of ≤10 prior to challenge.
* Non-smoker (no smoking within the last year and a history of less than 10 packs per year total) and agree to not use tobacco products during participation in the study.
* Female subjects of childbearing potential must:

  1. Not be breastfeeding
  2. Have a negative serum pregnancy test at screening and a negative urine pregnancy test on Day -1
  3. Will use oral, implantable, transdermal, or injectable contraceptives for 30 days prior to administration of the A/California/H1N1 2009 virus until the follow-up visit is performed.
  4. Use another reliable form of contraception approved by the Investigator (eg, intrauterine device, female condom, diaphragm with spermicide, cervical cap, use of condom by the sexual partner or a sterile sexual partner) from the time of screening until the follow-up visit is performed.
* Female subjects not of childbearing potential must:

  1. Be at least 1 year post-menopausal, or
  2. Be surgically sterile
* Male subjects able to father a child and sexually active with a female of childbearing potential, must agree to use a double barrier method of birth control (eg, condom with spermicidal foam, cream gel) and to not donate sperm during the study, from the day of enrollment until the Day 60 (±3) follow-up visit. If the female partner is using an effective method of contraception, a single barrier method of birth control for the male is acceptable.
* Comprehension of the study requirements, expressed availability for the required study period, and ability to be quarantined for up to 10 days and to attend the scheduled follow up visit.
* Negative alcohol and urine drug screening tests prior to entering quarantine.
* Being willing to adhere to the prohibitions and restrictions specified in this protocol

Exclusion Criteria:

* Prior receipt of any influenza vaccine within the previous 2 years.
* Significant adulthood history of seasonal hay fever or a seasonal allergic rhinitis or perennial allergic rhinitis or chronic or nasal or sinus condition such as chronic sinusitis.
* Abnormal nasal structure including septal deviation and nasal polyps, or surgery to the nose or nasopharynx within 6 months of signing the informed consent form or recent (within the last 6 months) history of frequent or prolonged episodes of epistaxis.
* Suffering from asthma, bronchiectasis, emphysema, chronic obstructive pulmonary disease or any other chronic lung disease. A history of childhood asthma before the age of 12 is acceptable provided the subject is asymptomatic without treatment. Subjects with a single episode of wheezing after age 12 (lasting less than 8 weeks) can be included at the investigator's discretion.
* A female who is pregnant or who is breast feeding
* Diastolic BP, systolic BP or, pulse not consistent with normal vital signs, based on investigator judgment.
* Current use or use of intranasal corticosteroids within the last 30 days prior to the administration of the investigational virus product (Study Day 1).
* Presence of significant uncontrolled medical, neurological or psychiatric illness (acute or chronic) as assessed by the Investigator. This includes, but is not limited to, institution of new surgical or medical treatment for a chronic condition), or a significant dose alteration for uncontrolled symptoms or drug toxicity within 3 months of screening and reconfirmed on Day -1 prior to challenge.
* Positive serology for HIV-1 or HIV-2, or HBsAg or HCV antibodies.
* Cancer or treatment for cancer, within 5 years, excluding basal cell carcinoma of the skin, which is allowed.
* Presence of immunosuppression or any medical condition that may be associated with impaired immune responsiveness, including, but not limited to, diabetes mellitus inflammatory bowel disease.
* Presently receiving (or history of receiving) or during the preceding 3-month period prior to screening, any medications or other treatments that may adversely affect the immune system such as allergy injections, immune globulin, interferon, immunomodulators, cytotoxic drugs or other drugs known to be frequently associated with significant major organ toxicity, or systemic corticosteroids (oral or injectable) azathioprine or mercaptopurine. Topical corticosteroids except intranasal will be allowed. Use of intranasal corticosteroids within the last 30 days prior to the administration of the investigational virus product (Study Day 1) is prohibited.
* Chronic condition requiring prescription or over-the-counter medicine, with the exception of vitamins.
* Anticipated presence of a household contact with documented severe immunosuppression (as defined by CD4 < 200/mm³ or an absolute neutrophil count < 1500/mm³), either as a result of disease and/or therapy.
* Anticipated presence of a household contact aged ≤ 5 years, aged > 64 years, or a pregnant contact within 2 weeks following challenge.
* Current professional activity as a caregiver or healthcare worker who will return to work within 2 weeks following challenge.
* History of anaphylactic type reaction to egg or egg protein, adverse reaction to oseltamivir, a previous severe allergic reaction with generalized uticaria, angioedema, or anaphylaxis
* History of Guillain-Barre syndrome
* History of drug or chemical abuse in the year before the study.
* Receipt of any investigational virus product or nonregistered drug within the 30 days prior to challenge or currently enrolled in any investigational drug study or intends to enroll in such a study within the ensuing study period.
* Receipt of blood or blood products 6 months prior to challenge or planned administration during the study period.
* Blood donation in the last 26 weeks.
* Acute disease within 72 hours prior to challenge, defined as the presence of a moderate or severe illness with or without fever (as determined by the Investigator through medical history and physical examination), or presence of a fever ≥ 38ºC oral.
* Elevated white cell count above 10.5 x 109/L or an absolute neutrophil count above 7.5 x 109/L.
* Any condition that, in the opinion of the Investigator, might interfere with the primary study objective.
* Drinks more than 1200 mL (or 5 cups of 240 mL per cup) of tea/coffee/cocoa/cola or other caffeinated beverage per day more than one day per week in the 2 weeks before screening.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2015-01-19 (Actual); Primary Completion 2015-08-10 (Actual); Study Completion 2015-08-10 (Actual)

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were enrolled at a single site in California
Pre-assignment Details: Enrolled participants with evidence of an infection, elevated blood pressure, or abnormal lab values prior to Day 1 did not receive the investigational virus product.
Groups:
- Cohort 1: 1:10 dilution of neat virus (0.25mL of 1:10 dilution per nostril of neat virus; approximate quantity 3.5 x 106TCID50/dose)
  Live, wild-type A/California/H1N1 2009 influenza virus
- Cohort 2: 1:5 dilution of neat virus (0.25mL of 1:5 dilution per nostril of neat virus; approximate quantity 7 x 106TCID50/dose)
  Live, wild-type A/California/H1N1 2009 influenza virus
- Cohort 3: 1:10 dilution of neat virus (0.5mL of 1:10 dilution per nostril of neat virus; approximate quantity 7 x 106TCID50/dose)
  Live, wild-type A/California/H1N1 2009 influenza virus
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Started | 12 | 11 | 12
Completed (All participants completed the influenza challenge, and 1 participant was lost in AE follow-up) | 11 | 11 | 12
Not Completed | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Total
Number analyzed (Participants) | 12 | 11 | 12 | 35
Age, Continuous [Median (Full Range); unit: years] | 38 [27 to 44] | 30 [23 to 43] | 29 [21 to 44] | 33 [21 to 44]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 4 | 15
  Male | 6 | 6 | 8 | 20
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 4 | 6 | 5 | 15
  Black or African American | 7 | 4 | 6 | 17
  Asian | 1 | 1 | 0 | 2
  Multiracial | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Viral Shedding
Description: Number of participants with viral shedding, assessed from nasopharyngeal swabs using RT-PCR and cell culture assay
Time Frame: Day 9
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 12 | 11 | 12
Participants
  Shedding | 8 | 4 | 7
  No Shedding | 4 | 7 | 5

2. Primary Outcome: Seroconversion
Description: Greater than or equal to 4-fold rise in HAI titer by study Day 60 relative to baseline
Time Frame: Day 60
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 11 | 11 | 12
Participants
  Less than 4-fold rise in HAI titer | 5 | 5 | 4
  Greater than or equal to 4-fold rise in HAI titer | 6 | 6 | 8

3. Secondary Outcome: Number and Severity of AEs
Description: The number of AEs in each Cohort rated as mild, moderate, or severe intensity
Time Frame: Day 60
Measure: Number; unit: events
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 11 | 11 | 12
events
  Mild | 9 | 3 | 2
  Moderate | 4 | 1 | 0
  Severe | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Participants were followed through Day 60 (±3) for adverse events.
Description: AEs were defined as any untoward medical occurrence whether or not considered related to the investigational virus product.
  The solicited signs and symptoms of influenza will not be reported as AEs as these constitute an endpoint of the study and will be recorded as such, unless a situation arises where it is the opinion of the Investigator to do so.
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/11 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/11 | 0/12
Other Adverse Events (participants affected / at risk) | 9/12 | 1/11 | 2/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=12) | Cohort 2 (N=11) | Cohort 3 (N=12)
Chest discomfort/tightness (General disorders) | 2 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 0 | 0
Headache (Nervous system disorders) | 2 | 0 | 0
Elevated liver enzymes (Renal and urinary disorders) | 2 | 0 | 0
Cold symptoms (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No